CLINICAL TRIAL: NCT01631747
Title: Maternal-Offspring Metabolics:Family Intervention Trial (MOMFIT)
Brief Title: Maternal-Offspring Metabolics:Family Intervention Trial
Acronym: MOMFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Linda Van Horn, Professor, Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK10-014; 1U01HL114344-01 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy; Weight Gain
Keywords: Pregnancy; Weight gain; Obesity; Pregnancy and weight gain
MeSH Terms: conditions — Weight Gain; Obesity; Gestational Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Group (Active Comparator): Mom and family continue their typical eating, activity and other lifestyle habits for 24 months. They are invited to attend quarterly classes addressing prenatal wellness and family topics.
  Interventions: Behavioral: Usual Care Group
- Lifestyle Intervention Group (Experimental): Women in the Intervention group will participate in a lifestyle program based on Moms'adopting a healthier diet and becoming more active for 24 months. Implementation is at approximately 15 weeks.Moms will meet individually with their Lifestyle Coach (LC)at least 3 times(more as needed, attend six sessions during pregnancy and one session after delivery. In addition moms will participate in monthly phone counseling sessions with Lifestyle Coach and complete daily tracking of diet & activity and use of pedometer
  Interventions: Behavioral: Lifestyle Intervention Group

INTERVENTIONS:
Behavioral: Lifestyle Intervention Group — Moms will meet individually with their Lifestyle Coach (LC)at least 3 times(more as needed, attend six sessions during pregnancy and one session after delivery. In addition moms will participate in monthly phone counseling sessions with Lifestyle Coach and complete daily tracking of diet & activity and use of pedometer
  Arms: Lifestyle Intervention Group
Behavioral: Usual Care Group — Mom and family continue their typical eating, activity and other lifestyle habits for 24 months. They are invited to attend quarterly classes addressing prenatal wellness and family topics.
  Arms: Usual Care Group

SUMMARY:
The prevalence of maternal overweight and obesity has nearly doubled in the United States since 1976. In 2004-2005, 42% of pregnant women had body mass index (BMI) above 25 versus 23% in 1993. Most American women are overweight/ obese (OW/OB) at conception, especially within certain racial, ethnic, and lower socioeconomic groups leading to increased adverse maternal and birth outcomes. This study will recruit, randomize and test in 300 ethnically diverse OW/OB pregnant women a behavioral intervention aimed at controlling gestational weight gain (GWG) through recommended diet, activity and lifestyle changes that are to be maintained postpartum. Outcomes include anthropometric (height, weight, percent body fat) metabolic (blood pressure, fasting glucose, insulin, HbA1c, lipids and C-reactive protein) and behavioral measures (diet. physical activity, sleep and stress). In addition, babies will be measured for length, weight and percent body fat. The goal is to limit excessive gestational weight gain through improved maternal lifestyle that can be maintained and modelled for the family post partum and beyond.

DETAILED DESCRIPTION:
A Randomized Control Trial is planned among ethnically diverse OW/OB pregnant women ages 18-45 years to be randomly assigned to the MOMFIT Active Intervention Group (AIG) or the Educational Control Group (ECG) plus standard obstetrical care. The Dietary Approaches to Stop Hypertension (DASH) diet, along with moderate physical activity and group intervention as utilized in the Diabetes Prevention Program (DPP), will be adapted for pregnant and postpartum women through individual visits to tailor calorie/nutrient/activity goals, plus group coaching sessions and electronic self-monitoring behavior. Evidence based motivational interviewing and state of the art self-monitoring tools involving the LoseIt app will be adapted for pregnant/postpartum women via smartphone or Internet access, along with tailored feedback and encouragement from the Lifestyle Coach. Prevention of excessive GWG and achievement of the Institute Of Medicine (IOM) weight gain goals will be compared between groups, whether ongoing adherence to the lifestyle interventions can be sustained through postpartum intervention. Approximately one third of the participants are expected to be minorities and/or from low income backgrounds. The primary outcome is gestational weight gain from baseline (self-reported prepregnancy weight) to near delivery (36 weeks) compared with IOM goals in both groups and postpartum weight retention between 6 weeks and 12 months postpartum. Additional outcome variables include changes in maternal Body Mass Index (BMI) and adiposity postpartum, blood pressure, blood glucose, insulin, Hemoglobin A1c (HbA1c), C-reactive Protein (CRP), and lipids, diet quality, and physical activity levels, offspring adiposity and anthropometrics, and glucose and C-peptide in cord blood

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Singleton viable pregnancy. A twin pregnancy reduced to singleton before 14 weeks by project gestational age. An ultrasound must be conducted before randomization that shows a fetal heartbeat; there should be no evidence of more than one fetus on the most recent pre-randomization ultrasound.
* Gestational age at randomization no earlier than 9 weeks 0 days and no later than 15 weeks 6 days based on an algorithm (see Section 3.4.3 below) that compares the last menstrual period (LMP) date and data from the earliest ultrasound
* Body mass index between 25-35 kg/m2 based on first trimester measured weight and on measured height. The earliest weight measurement before randomization, measured specifically for the study will be used.

Exclusion Criteria:

* In vitro fertilization (IVF) conception/ovulation induction w/ gonadotropins
* Weight gain of >15 pounds from reported prepregnancy weight to Baseline visit
* Current smoker
* Prior bariatric surgery
* In weight loss program w/in 3 months of conception
* History of alcohol or drug abuse within 5 years
* No access to internet and/or smartphone
* Unable to attend intervention/follow-up visits
* Unwilling/unable to commit to self-monitoring data collection
* Unable to complete intervention program
* Presence of any condition that limits walking or following diet recommendations
* Not fluent in English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2012-11; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda V Van Horn, PhD, Principal Investigator — Northwestern University; Alan Peaceman, MD, Principal Investigator — Northwestern Memorial Hospital
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital; Prentice Women's, Chicago, Illinois
  - Northwestern University: Dept of Preventive Medicine, Chicago, Illinois

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Van Horn L, Peaceman A, Kwasny M, Vincent E, Fought A, Josefson J, Spring B, Neff LM, Gernhofer N. Dietary Approaches to Stop Hypertension Diet and Activity to Limit Gestational Weight: Maternal Offspring Metabolics Family Intervention Trial, a Technology Enhanced Randomized Trial. Am J Prev Med. 2018 Nov;55(5):603-614. doi: 10.1016/j.amepre.2018.06.015. Epub 2018 Sep 24. PMID 30262148
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were screened from multiple practices at the Prentice Women's Hospital of Northwestern Memorial Hospital. Screening took place between Feb 2013-Dec 2015.
Pre-assignment Details: Women completed baseline clinic visit and two 24 hour recalls prior to randomization.
Groups:
- Lifestyle Intervention Group: Moms will meet individually with their Lifestyle Coach (LC)at least 3 times(more as needed, attend six sessions during pregnancy and one session after delivery. In addition moms will participate in monthly phone counseling sessions with Lifestyle Coach and complete daily tracking of diet & activity and use of pedometer
  Lifestyle Intervention Group: Women in the Intervention group will participate in a lifestyle program based on Moms'adopting a healthier diet and becoming more active for 24 months. Implementation is at approximately 15 weeks.Moms will meet individually with their Lifestyle Coach (LC)at least 3 times(more as needed, attend six sessions during pregnancy and one session after delivery. In addition moms will participate in monthly phone counseling sessions with Lifestyle Coach and complete daily tracking of diet & activity and use of pedometer
Period: Randomization Through End of Pregnancy
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Started | 141 | 140
Completed | 140 | 140
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Live Birth
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Started | 140 | 140
Completed | 136 | 139
Not Completed | 4 | 1
Not completed — Pregnancy Termination | 1 | 0
Not completed — MIscarriage | 2 | 0
Not completed — Stillbirth | 1 | 1
Period: One Year Infant Outcomes
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Started | 136 | 139
Completed | 123 | 130
Not Completed | 13 | 9
Not completed — Patient Refused | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Lifestyle Intervention Group | Total
Number analyzed (Participants) | 141 | 140 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (4) | 33 (4) | 33 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 140 | 281
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 30 | 60
  Not Hispanic or Latino | 111 | 110 | 221
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 20 | 34 | 54
  White | 99 | 79 | 178
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 141 | 140 | 281
Gestational Age at Randomization [Mean (Standard Deviation); unit: weeks] | 13 (1) | 13 (1) | 13 (1)
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg per meters-squared] | 31 (4) | 31 (4) | 31 (4)

OUTCOME MEASURES:

1. Primary Outcome: Gestational Weight Gain (GWG)
Description: The primary outcome is GWG as assessed continuously by the difference between the maternal weight measured at the baseline and at the 35-37 week visit.
Time Frame: 14-37 weeks
Population: Women who had at least one follow-up weight in addition to baseline clinic weight.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 140 | 140
kg | 12 (6) | 10 (6)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Sample size was based on an independent 2-sample t-test using a two-sided type 1 error rate of 0.05, and 80% power. Assuming a standard deviation (SD) of 15lbs (6.8kg), a clinically meaningful difference of 5lbs (2.4kg) between groups, and 10% attrition, a sample size of 150/group was required; Test type: Superiority; p = 0.01, t-test, 2 sided — p-value is not adjusted for multiple comparisons, and tested at an a priori type I error rate of 0.05
Statistical Analysis 2: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.02, Regression, Linear; adjusted for actual gestational age of 36 week weight, gestational age, bmi, and maternal age at randomization, maternal race and paternal race

2. Secondary Outcome: Percentage of Participants With Gestational Diabetes
Description: Oral Glucose Tolerance Test (OGTT) will be administered at 24-26wks, as part of routine obstetric visit. Difference in incidence of Gestational diabetes between study groups will be documented.
Time Frame: 24-26 weeks
Population: Inadequate testing was done for several participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 127 | 133
Participants | 9 | 7
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.54, Chi-squared

3. Secondary Outcome: Fasting Glucose
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 wks
Population: Participants with valid glucose measures
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 92 | 102
mg/dL
  Baseline | 87 [83 to 91] | 86 [82 to 90]
  35-37 Weeks | 85 [81 to 89] | 84 [80 to 89]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.89, t-test, 2 sided; T-test performed on change in glucose (log scale), but presented as Median and inter-quartile range for interpretability

4. Secondary Outcome: High-density Lipoprotein (HDL)
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 wks
Population: Participants with phlebotomy
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 94 | 106
mg/dL
  Baseline | 66 [58 to 78] | 71 [60 to 80]
  35-37 Weeks | 68 [57 to 79] | 70 [56 to 82]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.30, t-test, 2 sided; t-test performed on changes in HDL, but presented as median and IQR for ease of interpretation

5. Secondary Outcome: Low-density Lipoprotein (LDL)
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 weeks
Population: Participants with valid LDL measures
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 90 | 104
mg/dL
  Baseline | 95 [79 to 112] | 94 [78 to 117]
  35-37 Weeks | 146 [103 to 164] | 130 [106 to 163]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.69, t-test, 2 sided; t-test run on changes between groups. Data presented as median and IQR for ease of interpretation

6. Secondary Outcome: Total Cholesterol
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 Weeks
Population: participants with Phlebotomy at week 35
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 94 | 106
mg/dL
  Baseline | 188 [167 to 205] | 185 [164 to 208]
  35-37 Weeks | 255 [219 to 290] | 252 [222 to 281]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.19, t-test, 2 sided; t-test run on change between groups (log scale), but presented as median and IQR for ease of interpretation

7. Secondary Outcome: Triglycerides
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 Weeks
Population: Participants with phlebotomy at 35 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 94 | 106
mg/dL
  Baseline | 108 [86 to 138] | 109 [81 to 131]
  35-37 Weeks | 235 [187 to 300] | 223 [180 to 271]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.27, t-test, 2 sided; t-test used to compare changes between groups (log scale). Median and IQR are presented for ease of interpretation

8. Secondary Outcome: Leptin
Description: Blood will be collected at Baseline and 35-37 weeks.
Time Frame: 14-37 weeks
Population: Participants with phlebotomy at week 35
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 94 | 106
ug/L
  Baseline | 49 [40 to 58] | 50 [40 to 61]
  35-37 Weeks | 59 [49 to 68] | 54 [44 to 67]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.003, t-test, 2 sided; t-test performed on changes between groups (log scale). Median and IQR are presented for ease of interpretation

9. Secondary Outcome: Steady State Beta Cell Function
Description: Insulin resistance will be measured with the assistance of a computer program (HOMA Calculator v2.2.3, Diabetic Trial Unit, University of Oxford) which uses blood Glucose and Insulin measures to yield the Homeostatic Model Assessment (HOMA) Steady State beta cell function (%B). 100% is set at normal reference. Should not be interpreted alone, but in combination with Insulin Sensitivity (%S).
Time Frame: baseline (14 weeks) and 35-37 weeks
Population: Participants with valid glucose measures
Measure: Median (Inter-Quartile Range); unit: percentage of normal reference
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 92 | 102
percentage of normal reference
  Baseline | 120 [99 to 150] | 121 [98 to 145]
  35-37 Weeks | 174 [137 to 205] | 159 [133 to 195]
Statistical Analysis 1: Comparison: Usual Care Group; Test type: Superiority; p = 0.24, t-test, 2 sided; t-test run on change between groups (log scale), but presented as median and IQR for ease of interpretation

10. Secondary Outcome: Insulin Sensitivity
Description: Insulin resistance will be measured with the assistance of a computer program which will yield the Homeostatic Model Assessment (HOMA) Insulin Sensitivity (%S). 100% is equivalent to the normal reference, but needs to be interpreted in context of %B.
Time Frame: baseline(14 weeks) and 35-37 weeks
Population: Participants with valid glucose measures
Measure: Median (Inter-Quartile Range); unit: percentage of normal reference
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 92 | 102
percentage of normal reference
  Baseline | 78 [56 to 107] | 87 [59 to 112]
  35-37 Weeks | 51 [39 to 74] | 62 [41 to 80]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.32, t-test, 2 sided; t-test run on change between groups (log scale), but presented as median and IQR for ease of interpretation

11. Secondary Outcome: Insulin Resistance (IR)
Description: Insulin resistance will be measured with the assistance of a computer program (HOMA Calculator v2.2.3, Diabetic Trial Unit, University of Oxford) which uses blood Glucose and Insulin measures to yield the Homeostatic Model Assessment (HOMA) Insulin Resistance. HOMA IR (insulin resistance) is the reciprocal of insulin sensitivity (%S), as a percentage of a normal reference population (100/%S); Lower IR is better.
  Note: estimates are model-derived, and not linear approximations.
Time Frame: Baseline (14 weeks) and 35 weeks
Population: Participants with valid glucose levels.
Measure: Median (Inter-Quartile Range); unit: inverse proportion of normal reference
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 92 | 102
inverse proportion of normal reference
  Baseline | 1.3 [0.9 to 1.8] | 1.2 [0.9 to 1.7]
  35-37 Weeks | 2.0 [1.4 to 2.6] | 1.6 [1.3 to 2.4]
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.26, t-test, 2 sided; T-test performed on change between groups (log scale). Median and IQR are presented for ease of interpretation

12. Secondary Outcome: Birth Weight
Description: Neonatal Body measurements
Time Frame: Delivery
Population: Participants with live births
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 121 | 130
g | 3213 (524) | 3244 (489)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.62, t-test, 2 sided

13. Secondary Outcome: Birth Length
Description: Neonate birth measures
Time Frame: Delivery
Population: participants with live births
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 121 | 130
cm | 51 (3) | 51 (2)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.61, t-test, 2 sided

14. Secondary Outcome: Head Circumference
Description: Neonate birth measures
Time Frame: Delivery
Population: Live births
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 121 | 130
cm | 34 (2) | 34 (2)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.42, t-test, 2 sided

15. Secondary Outcome: Neonate Percent Body Fat
Description: Neonate percent body fat as measured by PeaPod, and air displacement plethysmography system.
Time Frame: Delivery
Population: Participants with PeaPod measurements
Measure: Mean (Standard Deviation); unit: percentage of weight
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 92 | 106
percentage of weight | 11.9 (4.2) | 11.2 (4.4)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.25, t-test, 2 sided

16. Secondary Outcome: Infant Weight
Description: Infant Body measurements
Time Frame: 1 year
Population: Participants with measured or reported 1 year infant weight
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 123 | 130
kg | 9.9 (1.2) | 9.9 (1.3)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.66, t-test, 2 sided

17. Secondary Outcome: Infant Length
Description: Infant body measurement
Time Frame: 1 year
Population: Participants with one year infant body measures
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Usual Care Group | Lifestyle Intervention Group
Number analyzed (Participants) | 118 | 125
cm | 76.3 (3.6) | 76.2 (3.5)
Statistical Analysis 1: Comparison: Usual Care Group vs Lifestyle Intervention Group; Test type: Superiority; p = 0.94, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Each participant was followed from initial contact through delivery for adverse events (approximately 7 months).
Arm/Group | Usual Care Group | Lifestyle Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/140
Serious Adverse Events (participants affected / at risk) | 29/141 | 18/140
Other Adverse Events (participants affected / at risk) | 5/141 | 3/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (N=141) | Lifestyle Intervention Group (N=140)
Pregnancy Loss/Termination (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) — Miscarriage, Termination, Antepartum stillbirth
Abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 — Placenta Abruption
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 6 (6) — Preeclampsia / severe preeclampsia / HELLP / eclampsia / high blood pressure
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1) — Cholestasis / elevated liver enzymes
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chorioamnionitis (Infections and infestations) | 1 (1) | 0 (0) — Intrapartum maternal infection
Vasa Previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Placenta Abnormality
Postpartum maternal infection (Surgical and medical procedures) | 1 (1) | 0 (0) — small bowel perforation
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — respiratory compromise
Congenital anomaly (Congenital, familial and genetic disorders) | 7 (7) | 2 (2) — Fetal Congenital anomaly; small centricular septal defects, pulmonary stenosis dysplastic pulmonary valve, trisomy 13, gastroschisis, esophagaeal atresia, trisomy 21, duodenal atresia.
NICU admission (General disorders) | 18 (18) | 12 (12) — Neonatal Intensive care unit admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (N=141) | Lifestyle Intervention Group (N=140)
Small for gestational age (Endocrine disorders) | 5 (5) | 3 (3) — Neonate born small for gestational age

LIMITATIONS AND CAVEATS:
The study recruited 281 participants, fewer than the target sample size of 300; this did not impact power for the primary outcome (higher retention rates), but requires attention when considering translational implications to a clinic setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT01631747/Prot_SAP_000.pdf